CLINICAL TRIAL: NCT04413123
Title: A Phase 2 Study of Cabozantinib in Combination With Nivolumab and Ipilimumab in Advanced Non-Clear Cell Renal Cell Carcinoma
Brief Title: Cabozantinib In Combo With NIVO + IPI In Advanced NCCRCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bradley A. McGregor, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Exelixis (Industry)
Responsible Party: Sponsor-Investigator, Bradley A. McGregor, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-789
Record Dates: First submitted 2020-03-26; First posted 2020-06-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Papillary Renal Cell Carcinoma; Unclassified Renal Cell Carcinoma; Translocation Renal Cell Carcinoma; Chromophobe Renal Cell Carcinoma; Collecting Duct Renal Cell Carcinoma; Renal Cell Carcinoma; Unresectable Advanced Renal Cell Carcinoma; Metastatic Ncc Renal Cell Carcinoma
Keywords: Papillary Renal Cell Carcinoma; Unclassified Renal Cell Carcinoma; Translocation Renal Cell Carcinoma; Chromophobe Renal Cell Carcinoma; Collecting duct Renal Cell Carcinoma; Renal Cell Carcinoma; Unresectable Advanced Renal Cell Carcinoma; Metastatic ncc Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Eligible patients will be enrolled and receive treatment with
  * Cycle 1-4 (cycles of 21 days)
    * Cabozantinib predetermined protocol dosage po daily
    * Nivolumab predetermined protocol dosage via IV every 3 weeks
    * Ipilimumab predetermined protocol dosage via IV every 3 weeks
  * After the first four cycles of therapy,
    * Cabozantinib determined protocol dosage po daily
    * Nivolumab predetermined protocol dosage via IV every 3 weeks (cycles of 28 days)
  Interventions: Drug: Cabozantinib; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib predetermined protocol dosage po daily
  Other Names: COMETRIQ™; CABOMETYX™
Drug: Nivolumab — Nivolumab predetermined protocol dosage via IV every 3 weeks
  Other Names: Opdivo®
Drug: Ipilimumab — Ipilimumab predetermined protocol dosage via IV every 3 weeks
  Other Names: Yervoy

SUMMARY:
This research study will assess whether cabozantinib, nivolumab and ipilimumab in combination are safe and effective in slowing down the growth of kidney cancer(renal cell carcinoma or RCC) that has advanced or spread to other areas the body.

DETAILED DESCRIPTION:
This research study involves an investigational drug combination not approved by the FDA (the U.S. Food and Drug Administration) for your kidney cancer.

The names of the study drugs in this investigational combination are:

* Cabozantinib
* Nivolumab
* Ipilimumab

The research study procedures include screening for eligibility, study treatment, participant evaluations and safety follow-up visits, in addition to general health status follow-up after study treatment.

It is expected that about 40 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed unresectable advanced or metastatic nccRCC, including but not limited to:

  * Papillary RCC, any type
  * Unclassified RCC
  * Translocation RCC
  * Chromophobe RCC
  * Collecting duct RCC
  * Renal cell carcinoma with 80% or more sarcomatoid features on primary nephrectomy specimen or a biopsy
  * Other nccRCC histologies in discussion with principal investigator
* Measurable disease as per RECIST 1.1. See Section 11 for the evaluation of measurable disease.
* Age ≥ 18 years
* ECOG performance status ≤1 (Karnofsky ≥70%, see Appendix A)
* Participants must undergo fresh tumor biopsy after registration but prior to the start of treatment unless medically unsafe or not feasible. If a fresh tumor biopsy is not medically safe or not feasible, confirmation of the availability of archival tumor tissue is required. For archival tissue, a recommended minimum of 20 unstained slides should be obtained.
* Normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥9g/dL (transfusions allowed)
  * total bilirubin ≤2.0 x institutional upper limit of normal with the following exception: patients with known Gilbert disease should have a serum bilirubin ≤ 3 x ULN
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal with the following exception: patients with known liver metastases should have AST and ALT ≤ 5 x ULN
* creatinine clearance ≥30 mL/min/1.73 m2 according to the Cockcroft-Gault equation.
* Normal coagulation INR ≤ 1.5
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 5 months after the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 7 months after completion of cabozantinib, nivolumab or ipilimumab administration.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

- Patients could be untreated or have received prior lines of therapies. Patients who receive prior therapy may receive only one VEGF based therapy. A combination therapy (e.g.

lenvatinib+everolimus) is considered 1 line of therapy.

* Previous therapy with CD137 agonists and immune checkpoint inhibitors, including but not limited to inhibitors of the PD-1/PD-L1 and/or CTLA-4 axes. Previous treatment with IFNα or IL-2 is allowed if received > 4 weeks from enrollment.
* Treatment with small molecule tyrosine kinase inhibitors within 2 weeks of enrollment, or any other anticancer agent within 4 weeks of enrollment.
* Prior therapy with cabozantinib
* Patients receiving any other therapeutic investigational agents.
* Treatment with hydroxychloroquine within two weeks of treatment start.
* Radiotherapy for nccRCC within 14 days of first study treatment with the exception of a single fraction of radiation administered for palliation of symptoms.
* Untreated brain metastases. Patients might be included if they underwent radiation therapy or surgery at least 4 weeks prior enrollment. Stability of the central nervous system disease should be confirmed by brain MRI or CT-scan or as determined by treating investigator. Patients should not be receiving prednisone dose >10 mg/d at C1D1.
* Other malignancy diagnosed within 2 years of first study treatment unless negligible risk of metastases or death (included but not limited to carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma, or other malignancy not deemed to impact patients 5-year life expectancy).
* Significant cardiovascular disorders including:

  * Significant cardiovascular disease including dyspnea of New York Heart Association (NYHA) class II or greater, myocardial infarction within the previous 3 months of first study treatment, unstable arrhythmias, unstable angina. Patients with known coronary artery disease or congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50%, must be on a stable and optimized in the opinion of the treating physician, in consultation with a cardiologist when appropriate.
  * Uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy is allowed.
  * Personal history of hypertensive crisis or hypertensive encephalopathy within the previous 3 months of registration.
  * Personal history of stroke or transient ischemic attack within 3 months of registration.
  * Significant vascular disease, such as but not limited to aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis, within 6 months of registration.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG). Furthermore, subjects with a history of additional risk factors for torsades de pointes (eg, long QT syndrome) are also excluded.
* Known history of severe allergic reactions attributed to compounds of similar chemical or biologic composition human antibodies, or known hypersensitivity to any component of cabozantinib, nivolumab or ipilimumab products.
* Systemic immunosuppressive medications including but not limited to: Corticosteroids at a dose > 10mg equivalent prednisone daily, cyclosporin, azathioprine, methotrexate, thalidomide, anti-tumor necrosis factor (TNF) agents, hydroxychloroquine, within 2 weeks of first study dose.

  * Patients who have received acute, low-dose systemic immunosuppressant medications may be enrolled.
  * Patients with adrenal insufficiency on physiologic replacement doses of steroids may be enrolled.
  * The use of inhaled, topical, intraocular, or intraarticular corticosteroids or mineralocorticoids are allowed
* Prior allogenic stem cell or solid organ transplant.
* Personal history of autoimmune disease including: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, type I diabetes mellitus, vasculitis, or glomerulonephritis. Patients with a history of autoimmune-related hypothyroidism on thyroid replacement hormone, or those with autoimmune dermatologic conditions not requiring the use of prednisone > 10 mg or equivalent are eligible.
* History of idiopathic pulmonary fibrosis, organized pneumonia, or evidence of active pneumonitis on screening imaging CT of the chest. History of radiation pneumonitis in the radiation field is permitted.
* History of following infectious diseases:

  * Active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening).
  * Active hepatitis C infection. Patients with positive hepatitis C antibody test are eligible if PCR is negative for hepatitis C viral DNA.
  * Infection requiring therapeutic oral or IV anti-microbials within 2 weeks of first study treatment. Patients receiving routine antimicrobial prophylaxis for dental procedures are eligible.
  * Known positive test for HIV.
* Administration of a live, attenuated vaccine within 3 weeks for first study treatment.
* Bleeding diathesis, or significant coagulopathy in the absence of therapeutic anticoagulation.
* Use of strong inhibitors and inducers of CYP3A4
* Significant bleeding, including but not limited to hematemesis, hematuria, hemoptysis of > 0.5 teaspoon (2.5 mL), within 3 months before registration.
* Invasion of major pulmonary blood vessels. A discussion with PI may be needed if invading lesions are suspected.
* Concomitant use of dipyramidole, ticlopidine, clopidogrel, cilostazol is excluded. Aspirin (≤ 325 mg per day) is allowed. Prophylactic anticoagulation with oral or parenteral anticoagulants for the patency of venous access devices or other indications is allowed.

Therapeutic use of low-molecular weight heparin (such as enoxaparin) and subcutaneous or oral Factor Xa inhibitors are allowed. Use of warfarin is prohibited.

* Significant GI conditions at risk of perforation or bleeding, including but not limited to:

  * Active GI obstruction or requirement of routine parenteral nutrition or tube feedings.
  * Personal history of abdominal or tracheoesophageal fistula or GI perforation within 6 months of registration.
  * Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
  * Serious, non-healing or dehiscing wound or active ulcer.
* Major surgical procedure to include major dental, oral or maxillofacial procedures within 14 days of first study treatment.
* Proteinuria as demonstrated by > 1.5 gram of protein in a 24-hour urine collection. All patients with ≥ 2+ protein on urinalysis must undergo 24-hour urine collection for protein.
* Unable to swallow pills.
* Malabsorption syndrome.
* Inability to receive IV medications
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | tart of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started up to 21 Months
  Percent of patients who achieve overall response (CR or PR) by RECIST 1.1 will be summarized with 80% two-sided exact binomial confidence intervals (CI)

SECONDARY OUTCOMES:
Duration of response (DOR) | first documentation of response, to the earlier of the first documentation of disease progression or death from any cause, and calculated for patients with a best confirmed response of CR up to 21 Months
  will be estimated using the method of Kaplan-Meier, for all patients and by histology subtypes. M
Progression-free survival (PFS) | trial treatment start to the earlier of progression or death due to any cause per investigator assessment. Participants alive without disease progression are censored at date of last disease evaluation up to 21 Months
  the method of Kaplan-Meier, for all patients and by histology subtypes evaluation.
Overall survival (OS) | from trial treatment start to death due to any cause or censored at date last known alive up to 21 Months
  the method of Kaplan-Meier, for all patients and by histology subtypes
"Number of Participants with TreatmentRelated Adverse Events as Assessed by CTCAE version 5. | Baseline, day 1 of every cycle (21 days for first 4 cycles and then 28 days for each cycle tehreafter) and End of Treatment up 21 months
  For toxicity reporting, all adverse events will be graded and analyzed using CTCAE version 5.
Quality of life- FKSI-19 Scale | 12 weeks for the first assessment, then every 8 weeks (+/- 7 days) for the first 6 months. Then take place every 12 weeks (+/- 7 days)
  The Functional Assessment of Cancer Therapy-Kidney Symptom (FKSI-19) is a 19 item questionnaire with each item scored on a scale of 0-4 for a total score of 0-76 with higher scores indicating fewer symptom
Quality of life-BFI Questionaire | 2 weeks for the first assessment, then every 8 weeks (+/- 7 days) for the first 6 months. Then take place every 12 weeks (+/- 7 days)
  The Brief Fatigue Inventory (BFI) is a 9-item questionnaire with each item scored on a scale of 0-10.
  Scores are categorized as mild (1-3), moderate (4-6), or severe (7-10). A global fatigue score can be found by averaging the score obtained on each test item completed
Objective response rate (ORR) | defined as the percentage of patients with partial (PR) or complete response (CR) as best overall response according to RECIST 1.1 by investigator assessment up to 21 Months
  ORR by RECIST 1.1 according to histology subtypes (Papillary RCC versus other histology types) will be summarized with 80% two-sided exact CIs.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley McGregor, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham & Woman's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - UT Southwestern Medical, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu